CLINICAL TRIAL: NCT01272076
Title: Cirrus HD-OCT Measurement of Area of Increased Light Penetration Under the Retinal Pigment Epithelium (RPE)
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD-OCT-GA-2010-1-v2
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-12

CONDITIONS: Age Related Macular Degeneration; Geographic Atrophy
Keywords: Age Related Macular Degeneration; Geographic Atrophy; Imaging; OCT
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dry AMD and geographic atrophy: Patients diagnosed with dry AMD and geographic atrophy

SUMMARY:
The objective of this study is to compare Cirrus HD-OCT automated measurements of the illumination area under the retinal pigment epithelium (RPE) to expert manual measurements of areas of hypofluorescence typical of geographic atrophy in fundus autofluorescence (FAF) images.

DETAILED DESCRIPTION:
Specific Objectives:

1. To compare Cirrus HD-OCT automated measurements of the illumination area under the RPE to expert manual measurements of areas of hypofluorescence typical of geographic atrophy in fundus autofluorescence (FAF) images.
2. To describe the differences and similarities between Cirrus HD-OCT and fundus autofluorescence images of subjects with geographic atrophy secondary to dry age-related macular degeneration (AMD).
3. To determine the clinical factors that affect the Cirrus HD-OCT automated measurements of the illumination area under the RPE.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 50 years of age and older diagnosed to have advanced dry AMD with geographic atrophy.
* Geographic atrophy lesions should:

  * Not be greater than 5 mm at the widest diameter. The entire lesion(s) should fit into the 6x6 mm scan area of the Cirrus HD-OCT.
  * Not be smaller than 1.25 mm2.
  * Not be confluent with peri-papillary atrophy.
  * Not be combined with other lesions such as CNVs.
* Able and willing to make the required study visit.
* Able and willing to give consent and follow study instructions.

Exclusion Criteria:

* History of retinal surgery, laser photocoagulation, and/or radiation therapy to the eye.
* Evidence of other retinal diseases of the eye, including wet AMD, diabetic retinopathy, diabetic macular edema, or significant vitreomacular traction upon dilated examination, or upon evaluation of retinal photos.
* Thick media opacity or inability to fixate that precludes obtaining acceptable scans.
* Concomitant use of hydrochloroquine and chloroquine.
* Unable to make the required study visit.
* Unable to give consent or follow study instructions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelina M Gordon, MD, Principal Investigator — TLC Eye Care and Laser Center; Eugene S Lit, M.D., Principal Investigator — East Bay Retina Consultants
Locations (2):
- United States (2):
  - East Bay Retina Consultants, Inc., Oakland, California
  - TLC Eyecare and Laser Centers, Jackson, Michigan

REFERENCES:
- [Background] Schmitz-Valckenberg S, Fleckenstein M, Scholl HP, Holz FG. Fundus autofluorescence and progression of age-related macular degeneration. Surv Ophthalmol. 2009 Jan-Feb;54(1):96-117. doi: 10.1016/j.survophthal.2008.10.004. PMID 19171212
- [Background] Holz FG, Bindewald-Wittich A, Fleckenstein M, Dreyhaupt J, Scholl HP, Schmitz-Valckenberg S; FAM-Study Group. Progression of geographic atrophy and impact of fundus autofluorescence patterns in age-related macular degeneration. Am J Ophthalmol. 2007 Mar;143(3):463-72. doi: 10.1016/j.ajo.2006.11.041. Epub 2006 Dec 22. PMID 17239336
- [Background] Hwang JC, Chan JW, Chang S, Smith RT. Predictive value of fundus autofluorescence for development of geographic atrophy in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2006 Jun;47(6):2655-61. doi: 10.1167/iovs.05-1027. PMID 16723483
- [Background] Lujan BJ, Rosenfeld PJ, Gregori G, Wang F, Knighton RW, Feuer WJ, Puliafito CA. Spectral domain optical coherence tomographic imaging of geographic atrophy. Ophthalmic Surg Lasers Imaging. 2009 Mar-Apr;40(2):96-101. doi: 10.3928/15428877-20090301-16. PMID 19320296
- [Background] Sunness JS, Margalit E, Srikumaran D, Applegate CA, Tian Y, Perry D, Hawkins BS, Bressler NM. The long-term natural history of geographic atrophy from age-related macular degeneration: enlargement of atrophy and implications for interventional clinical trials. Ophthalmology. 2007 Feb;114(2):271-7. doi: 10.1016/j.ophtha.2006.09.016. PMID 17270676
- [Background] Yehoshua Z, Rosenfeld PJ, Gregori G, Feuer WJ, Falcao M, Lujan BJ, Puliafito C. Progression of geographic atrophy in age-related macular degeneration imaged with spectral domain optical coherence tomography. Ophthalmology. 2011 Apr;118(4):679-86. doi: 10.1016/j.ophtha.2010.08.018. Epub 2010 Oct 29. PMID 21035861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 subjects were enrolled between 1/10/2011 - 2/25/2011. The study was conducted at Retina Specialist clinics.
Pre-assignment Details: After enrollment a screening image of the retina is done to ensure that the area of Geographic Atrophy is consistent with the inclusion criteria. We enrolled 85 subjects, however, 19 were determined not to be eligible per study protocol. In addition, images of 14 subjects did not meet predetermined qualification criteria per study protocol.
Groups:
- Dry AMD With Geographic Atrophy: Patients diagnosed with dry AMD and geographic atrophy
Period: Overall Study
Arm/Group | Dry AMD With Geographic Atrophy
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GA Group: Patients diagnosed with dry AMD and geographic atrophy
Arm/Group | GA Group
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Difference in mm Squared of Cirrus HD-OCT Automated Measurements of the Illumination Areaa Under the RPE to Expert Manual Measurement of Areas of Hypofluorescence Typical of Geographic Atrophy (GA).
Description: In retinal areas with atrophy, light emitted from the Cirrus penetrates the sclera and choroid which are more reflecting compared with the Retinal Pigment Epithelium (RPE). The areas with higher illumination are associated with areas of Geographic Atrophy (GA), and allow to quantify how big is the area of atrophy. The study will assess the difference between Cirrus HD-OCT measurements of areas of increased illumination under the RPE to hypofluorescence areas on fundus photos as assessed manually by retina specialists.
Time Frame: August 2011
Population: Subjects with dry AMD and Geographic Atrophy. The required sample size was calculated based on previous experience with the device and its variability.
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- GA Group: Inter-device variability in measuring the area of Geographic Atrophy. 3 acceptable scans from 3 Cirrus HD-OCT devices (total of 9) were taken by one operator in this phase.
Arm/Group | GA Group
Number analyzed (Participants) | 52
mm^2 | 0.1 (1.9)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the entire period of the study.
Groups:
- GA Group: Patients with dry age related macular degeneration and geographic atrophy.
Arm/Group | GA Group
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

LIMITATIONS AND CAVEATS:
No adverse event were found or reported for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results until the device is released on the market.